CLINICAL TRIAL: NCT00401648
Title: A Placebo-controlled, Single-blind, Multi-center Study to Explore the Photoparoxysmal Response in Photosensitive Epileptic Subjects After One Single Oral Dose of Brivaracetam in Capsules.
Brief Title: Effect of Brivaracetam in Photosensitive Epileptic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: N01069; Protocol Number RPCE02D2304
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Epilepsy
Keywords: POC; photosensitive; epileptic; brivaracetam; PPR; AED
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

INTERVENTIONS:
Drug: Brivaracetam

SUMMARY:
to assess the effect of brivaracetam on the photoparoxysmal EEG response in photosensitive epileptic subjects

ELIGIBILITY:
Inclusion Criteria:

* epileptic subjects with generalized PPR

Exclusion Criteria:

* more than 2 concomitant antiepileptic drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2002-09; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Identify lowest single oral dose producing maximal decrease or suppression of intermittent photic stimulation (IPS)photoparoxysmal response (PPR) in photosensitive epileptic subjects pre-dose
post placebo during 24h and post brivaracetam for up to 72 h

SECONDARY OUTCOMES:
Assess relationship between plasma concentrations and changes in photosensitivity frequency range, time of onset and duration of suppressing effect
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Philipp von Rosenstiel, MD., Study Director — UCB Pharma
Locations (5):
- France (4):
  - Marseille
  - Paris
  - Rouen
  - Strasbourg
- Kork, Germany